CLINICAL TRIAL: NCT02722382
Title: Putting Patients at the Center of Kidney Care Transitions
Brief Title: Putting Patients at the Center of Kidney Care Transitions (PREPARE NOW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Geisinger Clinic (Other); Johns Hopkins University (Other); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00074588
Record Dates: First submitted 2016-03-17; First posted 2016-03-30 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Nephrology Care (No Intervention): Nephrology care at Geisinger Health System.
- Patient-Centered Kidney Transitions Care (Active Comparator): Health system intervention which will implement informatics tools (including a disease registry, predictive modeling, and advance directives) and a disease specific care manager who will provide services and navigate patients through kidney disease transitions.
  Interventions: Other: Patient-Centered Kidney Transitions Care

INTERVENTIONS:
Other: Patient-Centered Kidney Transitions Care — In a multi-faceted pragmatic approach, the intervention will 1) implement new electronic health information tools to help providers recognize patents in need of Kidney Transitions Care and focus their attention on patients' values and treatment preferences; and 2) implement a Kidney Transitions Specialist who will provide and facilitate integrated delivery of patient support programs that provide patients with knowledge, skills, and assistance to manage their disease, make high-quality treatment decisions, obtain needed psychosocial support, and navigate complex treatment plans.
  Other Names: PREPARE NOW
  Arms: Patient-Centered Kidney Transitions Care

SUMMARY:
Objective: The investigators will change the health system to improve care patients receive as they transition through earlier stages of kidney disease toward kidney failure. They will study whether these changes lead to patients' improved health and well-being.

Methods: The investigators will conduct this study in Geisinger Health System kidney specialty clinics. The study will implement 'Patient Centered Kidney Transitions Care' which will (1) give doctors tools to help them recognize when patients should prepare for kidney failure and help them support patients' early and informed treatment decisions; and (2) add a 'Kidney Transitions Specialist' to the health care team to help patients learn about kidney disease, learn self-care skills, make informed decisions, get psychosocial support, and coordinate their care. Four (4) clinics will be randomly assigned to provide Patient Centered Kidney Transitions Care, and four (4) to provide their usual care. The investigators will study differences in patients' outcomes among those treated in clinics providing Patient Centered Kidney Transitions Care compared to those treated in clinics providing usual care.

Patient Outcomes: Patients have told us they want to have 'control' over their disease transitions and to have the best quality of life possible. The investigators will measure patients' empowerment, confidence with their self-care, their decisions to start self-care treatments for kidney failure, and their hospitalizations. They will also measure whether doctors record patients' treatment preferences in the medical record before patients develop kidney failure.

Patient and Stakeholder Engagement: This study responds to reports from hundreds of patients and caregivers who want better care. Patients and caregivers from around the US are part of our investigative team, and they will participate in all aspects of our study. The investigators are also engaging key stakeholders in the kidney community, including patients, providers, payers, and regulators.

Anticipated Impact: If effective, Patient Centered Kidney Transitions Care will provide a model of care can improve the lives of patients and families with kidney disease across the US.

DETAILED DESCRIPTION:
Background and Significance

Chronic kidney disease affects 20 million US adults who experience multifold excess morbidity and mortality compared to the general public. Over 115,000 patients develop kidney failure each year. For these patients, disease is often accompanied by unpredictable rapid rates of kidney function decline in its later stages. Unpredictable declines in kidney function commonly result in poorly planned transitions from seemingly stable chronic disease management to urgent or emergent needs for kidney failure treatments. These sudden transitions are often medically and psychologically traumatic for patients. Without advance planning and support, most patients initiate dialysis emergently, and they are unprepared to undergo substantial life changes and disability associated with treatments such as thrice-weekly hemodialysis. They also miss important early opportunities to select treatments (e.g., self care dialysis at home or kidney transplants) that could align with their values and improve their health.

Since it is difficult to predict who will suddenly develop kidney failure, all patients with later stage CKD should (a) be equipped to manage risks for disease progression and (b) learn about treatment options for kidney failure with enough time to understand and plan for possible treatments. Plans for some treatments, such as kidney transplant, are complex, requiring multiple referrals, diagnostic tests, and medical visits. The loss of kidney function is also, in some cases, accompanied by cognitive decline or by emotional disturbances (including denial, fear, or depression). As a result, patients need time to assimilate information and support to help them make informed decisions, coordinate their care, and obtain psychosocial help.

Health system support for patients' kidney disease transitions is often inadequate. As a result, patients have poor understanding of kidney disease treatments, feel care is not patient centered, and are 'blind-sided' by the seemingly catastrophic initiation of dialysis-- causing suffering and receipt of treatments they don't want. Efficacious educational, psychosocial, and care management interventions exist, but they are implemented in piecemeal fashion and are not readily accessible. Health system infrastructure and resources enabling integrated delivery of efficacious interventions may be the crucial missing link to ensuring patients' are supported through their to kidney failure and to improving their health and well-being.

Study Aims

The investigators seek to improve health systems' capacities to provide comprehensive care for patients as they transition from chronic kidney disease to kidney failure. Specifically, they will:

1. Establish a Patient Centered Kidney Transitions Care infrastructure that (a) prioritizes kidney patients' informed self-care and treatment decisions and (b) supports patients through their transitions across kidney disease stages by providing education, psychosocial support, and biomedical preparation
2. Study the effectiveness of the new Patient Centered Kidney Transitions Care infrastructure to improve patients' values-aligned kidney care, empowerment, and well-being

Study Description

The investigators will perform a cluster randomized controlled trial among 8 nephrology clinics in Geisinger Health System. Clinics provide nephrology care for over 2.6 million patients in 44 rural and suburban counties in eastern Pennsylvania. The study will target adults (age >18 years) with estimated glomerular filtration rates of <30 ml/min/1.73m2 or increased risk of disease progression. Practice populations are substantially rural with moderate to low education and advanced age. Practices serve 997 patients, and we anticipate 498 patients in each arm (each arm comprised of 4 practices).

In four clinics, the investigators will implement 'Patient Centered Kidney Transitions Care'. This intervention will implement two major health system changes, including (1) new electronic health information tools to alert providers when patients need kidney transitions care and to help them establish patients' preference aligned care; and (2) add a 'Kidney Transitions Specialist' to the health care team plus resources to support patients' transitions. Electronic health information tools will include (a) a disease registry and personalized risk prediction tools to prompt physicians when patients need transitions support and prepare patients for kidney failure when the time is right, and (b) a modular computer application which will help patients enter their values and treatment preferences into their own health records and help providers track their care. The Kidney Transitions Specialist will (1) facilitate patients' education and engage in shared decision-making with patients and caregivers; (2) empower patients to improve self-care through behavioral training; (3) engage peer and professional social and emotional support; (4) navigate patients through multi-step biomedical plans; and (5) advocate for aligning patients' care with their values. We will compare outcomes in clinics implementing Patient Centered Kidney Transitions Care to outcomes in four clinics that will proceed with routine nephrology care, which does not include health information tools or changes to the health care team or programs.

Primary outcomes will measure patients' empowerment, self-efficacy with self-care, decisions to start self-care treatments, and hospitalizations. The investigators will also measure documentation of patients' preferences in the electronic health record. These outcomes were chosen because patients have told us they want to feel they have 'control' over their disease and they want the best quality of life possible.

Long term, these findings will provide important information on how to improve the health and well being of patients as they transition from chronic kidney disease to kidney failure. If effective, this work will provide a model that can be replicated by health systems across the US.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving care at Geisinger nephrology practices
* Age 18 and older
* Advanced Kidney disease (determined by estimated glomerular filtration rates (eGFR) or presence of albuminuria)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1572 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in % patients feeling in control of their decision-making | Baseline, 36 months
  Change in % patients feeling in control of their decision-making
Change in number of Hospitalizations | Baseline, 36 months
  Change in number of Hospitalizations
Change in % patients with advance directives for kidney care | Baseline, 36 months
  Change in % patients with advance directives for kidney care

SECONDARY OUTCOMES:
Change in % self-care patients with biomedical care plans | Baseline, 36 months
  Change in % self-care patients with biomedical care plans
Change in % patients with values aligned care | Baseline, 36 months
  Change in % patients with values aligned care
Change in % patients with preferences for renal replacement therapy documented | Baseline, 36 months
  Change in % patients with preferences for renal replacement therapy
Change in % patients with emergency dialysis initiation | Baseline, 36 months
  Change in % patients with emergency dialysis initiation
Change in months to kidney failure | Baseline, 36 months
  Change in months to kidney failure
Change in % patients with vascular access (e.g., fistula) in place at dialysis initiation | 36 months
  Change in % patients with vascular access (e.g., fistula) in place at dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Leigh E Boulware, MD, Principal Investigator — Duke University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Browne T, Jones S, Cabacungan AN, Lang-Lindsey K, Schmidt L, Jackson G, Schatell D, Damron KC, Ephraim PL, Hill-Briggs F, Bolden S, Swoboda A, Ruff S, Danielson P, Littlewood D, Singer D, Stewart S, Vinson B, Clynes D, Green JA, Strigo TS, Boulware LE. The Impact of COVID-19 on Patient, Family Member, and Stakeholder Research Engagement: Insights from the PREPARE NOW Study. J Gen Intern Med. 2022 Apr;37(Suppl 1):64-72. doi: 10.1007/s11606-021-07077-w. Epub 2022 Mar 29. PMID 35349019
- [Derived] Green JA, Ephraim PL, Hill-Briggs F, Browne T, Strigo TS, Hauer CL, Yule C, Stametz RA, Littlewood D, Pendergast JF, Peskoe S, Clair Russell JS, Norfolk E, Bucaloiu ID, Kethireddy S, Davis D, dePrisco J, Malloy D, Fulmer S, Martin J, Schatell D, Tangri N, Sees A, Siegrist C, Breed J Jr, Billet J, Hackenberg M, Bhavsar NA, Boulware LE. Integrated Digital Health System Tools to Support Decision Making and Treatment Preparation in CKD: The PREPARE NOW Study. Kidney Med. 2021 May 24;3(4):565-575.e1. doi: 10.1016/j.xkme.2021.03.009. eCollection 2021 Jul-Aug. PMID 34401724
- [Derived] Browne T, Swoboda A, Ephraim PL, Lang-Lindsey K, Green JA, Hill-Briggs F, Jackson GL, Ruff S, Schmidt L, Woods P, Danielson P, Bolden S, Bankes B, Hauer C, Strigo T, Boulware LE. Engaging patients and family members to design and implement patient-centered kidney disease research. Res Involv Engagem. 2020 Nov 1;6(1):66. doi: 10.1186/s40900-020-00237-y. PMID 33292683
- [Derived] Green JA, Ephraim PL, Hill-Briggs FF, Browne T, Strigo TS, Hauer CL, Stametz RA, Darer JD, Patel UD, Lang-Lindsey K, Bankes BL, Bolden SA, Danielson P, Ruff S, Schmidt L, Swoboda A, Woods P, Vinson B, Littlewood D, Jackson G, Pendergast JF, St Clair Russell J, Collins K, Norfolk E, Bucaloiu ID, Kethireddy S, Collins C, Davis D, dePrisco J, Malloy D, Diamantidis CJ, Fulmer S, Martin J, Schatell D, Tangri N, Sees A, Siegrist C, Breed J Jr, Medley A, Graboski E, Billet J, Hackenberg M, Singer D, Stewart S, Alkon A, Bhavsar NA, Lewis-Boyer L, Martz C, Yule C, Greer RC, Saunders M, Cameron B, Boulware LE. Putting patients at the center of kidney care transitions: PREPARE NOW, a cluster randomized controlled trial. Contemp Clin Trials. 2018 Oct;73:98-110. doi: 10.1016/j.cct.2018.09.004. Epub 2018 Sep 12. PMID 30218818
- [Derived] Yee J. Improving Transitions in CKD: Failure Mode. Adv Chronic Kidney Dis. 2016 Jul;23(4):211-4. doi: 10.1053/j.ackd.2016.05.001. No abstract available. PMID 27324671